CLINICAL TRIAL: NCT00188136
Title: Phase II Study of Early Allogeneic Blood Stem Cell Transplantation During Induction-chemotherapy Induced Aplasia in High-risk Acute Myeloid Leukemia
Brief Title: Early Allogeneic Blood Stem Cell Transplantation in High-risk Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Carl Gustav Carus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDEATX
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML, allogeneic transplantation, high-risk, karyotype
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Melphalan; fludarabine

INTERVENTIONS:
Drug: Melphalan, ATG, Fludarabine — allo Tx during aplasia

SUMMARY:
Karyotype is a major prognostic risk factor in patients with acute myeloid leukemia (AML) translating into unfavourable outcome in case of poor-risk cytogenetic aberrations. Several studies have shown that allogeneic hematopoietic stem cell transplantation (HSCT) after myeloablative conditioning rather than autologous HSCT or consolidation chemotherapy result in long-term disease control in this group of patients when achieving a first complete remission. Nevertheless, the complete remission rate achievable is significantly lower than in patients with a more favourable risk profile. In fact, only the minority of AML patients with poor-risk cytogenetics, although having a suitable donor, proceed to HSCT due to refractory disease or infectious complications during induction chemotherapy (IC). Further, new data show that the course of therapy can be estimated as early as two weeks after the initiation of the first course of IC with patients presenting with more than 10 % marrow blasts doing significantly worse than those with a better clearance of blasts. As a result, the chance to obtain a durable remission is considerably low and most patients with bad-risk cytogenetics or failure to achieve blast clearance do not proceed to an allogeneic approach. Together these data indicate that early treatment intensification is warranted in order to provide the potential curative benefit of allogeneic HSCT to the majority of high-risk AML patients.

We have shown that reduced-intensity conditioning (RIC) followed by allogeneic PBSC applied during aplasia after the first cycle of IC in newly-diagnosed high-risk AML patients is feasible and can result in a sustained disease control. These data prompted us to further evaluate in a prospective trial an early "up-front HSCT" in patients with newly-diagnosed high-risk AML defined by karyotype and insufficient blast clearance after the first cycle of IC.

The goal was to provide an allogeneic HSCT as early as possible after diagnosis in AML patients.

DETAILED DESCRIPTION:
Only patients with newly-diagnosed AML are eligible for this prospective study. An immediate donor-search, either within the family or in volunteer donor registries, will be performed at diagnosis irrespective of the expected risk profile. All patients will receiv at least one cycle of IC. Inclusion criteria for early allogeneic transplantation are either poor risk cytogenetics and/or bad response to the first cycle of IC defined by more than 10% marrow blasts on day 15. If a patient meets one of those criteria they could enter the early allogeneic HSCT trial after providing informed consent. DNA-based HLA-typing of donor and recipient will be performed using high resolution (4 digits) for HLA - A, B, DRB1 and DQB1 and intermediate resolution (2 digits) for HLA- C.

During IC-induced aplasia after the 1st or 2nd cycle a fludarabine-based reduced intensity conditioning therapy will be started if a donor is available. All patients receive fludarabine 30 mg/m2 i.v. daily for five days (day- 6 to -2) and melphalan 150 mg/m² on day-2. Antithymocyte globulin (ATG Fresenius 10 mg/kg/day day -5 to -2, total dose 40 mg/kg, Fresenius, Bad Homburg, Germany) will be applied after transplantation from unrelated or HLA mismatched family donors. PBSC grafts will be preferred. As immunosuppression cyclosporin A (CsA) is either administered intravenously at a dose of 3 mg/kg/day or given at an bioequivalent amount of the oral formulation in two divided doses starting on the day before blood stem cell infusion (day -1). The dose of CsA is adjusted to maintain blood levels between 150 and 250 ng/ml. Starting on day 50, oral CsA administration will be tapered by 5% weekly if GVHD was inactive. Acute and chronic GvHD will be treated with prednisone, CsA or tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* newly-diagnosed AML
* either poor risk cytogenetics and/or bad response to the first cycle of IC defined by more than 10% marrow blasts on day 15
* HLA-compatible donor (maximum one HLA-antigen mismatch)

Exclusion Criteria:

* no donor
* Age < 16 years > 75 years
* Cardiac insufficiency requiring treatment or symptomatic coronary artery disease
* Hepatic disease, with AST > 2 times normal
* Severe hypoxemia , pO2 < 70 mm Hg, with decreased DLCO < 70% of predicted; or mild hypoxemia, pO2 < 80 mm Hg with severely decreased DLCO < 60% of predicted
* Impaired renal function (creatinine > 2 times normal or creatinine clearance < 50% for age, weight, height)
* HIV-positive patients due to risk of reactivation or acceleration of HIV replication
* Female patients who are pregnant or breast feeding due to risks to fetus from conditioning regimen and potential risks to nursing infants
* Life expectancy severely limited by diseases other than malignancy

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-08; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Total and relapse-free survival rate one year after the stem cell transplantation | 5 years

SECONDARY OUTCOMES:
Incidence of acute GvHD | 100 days
Safety (evaluated after Common Terminology Criteria for Adverse Events [CTCAE] v 3.0) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bornhauser, Prof, Principal Investigator — University hospital Carl Gustav Carus Dresden
Locations (1):
- University hospital Carl Gustav Carus, Dresden, Germany

REFERENCES:
- [Result] Platzbecker U, Thiede C, Freiberg-Richter J, Rollig C, Helwig A, Schakel U, Mohr B, Schaich M, Ehninger G, Bornhauser M. Early allogeneic blood stem cell transplantation after modified conditioning therapy during marrow aplasia: stable remission in high-risk acute myeloid leukemia. Bone Marrow Transplant. 2001 Mar;27(5):543-6. doi: 10.1038/sj.bmt.1702819. PMID 11313690